CLINICAL TRIAL: NCT03559309
Title: A Pilot Study Investigating the Effects of Lipid-therapy Intensification With Alirocumab on Endothelial Function, Carotid Arteries, Lipoprotein Particle Subfractions, Inflammation and Post-prandial Lipemia in Clinical Routine
Brief Title: Investigating the Effects of Lipid-therapy Intensification With Alirocumab on Endothelial Function, Carotid Arteries, Lipoprotein Particle Subfractions, Inflammation and Post-prandial Lipemia
Acronym: ALIROCKS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19 Pandemic Measures
Sponsor: Medical University of Graz (Other)
Collaborators: numares AG (Unknown); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ALIROCKS_05MAR2018_V3
Record Dates: First submitted 2018-05-22; First posted 2018-06-18 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Atherosclerosis; Hypercholesterolemia; Post Prandial Lipemia; Cardiovascular Diseases
MeSH Terms: conditions — Atherosclerosis; Hypercholesterolemia; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Alirocumab (Other): Medical Treatment (Clinical Routine)
  Interventions: Diagnostic Test: Magnet Resonance Tomography, Carotid Arteries Sonography, Flow-mediated Dilation, Fat-tolerance Test, Laboratory Testing

INTERVENTIONS:
Diagnostic Test: Magnet Resonance Tomography, Carotid Arteries Sonography, Flow-mediated Dilation, Fat-tolerance Test, Laboratory Testing — Patients treated with Alirocumab in the clinical routine will have additional diagnostic tests as stated above. The clinical trial will be conducted as an open label, single arm study. The diagnostic tests will be done at baseline (BL) and after 10 weeks of treatment (W10) with Alirocumab.

SUMMARY:
A prospective, open-label, pilot study with 24 cardiovascular high risk patients (N=24) having insufficient Low density lipoprotein cholesterin (LDL-C) reduction despite standard of care lipid-modifying therapies (LMTs), to evaluate the effects of potent lipid-therapy intensification via the recently approved monoclonal, human anti-PCSK9 antibody Alirocumab on endothelial function, inflammation, lipoprotein particle subfractions, carotid arteries and post-prandial lipemia in clinical routine at the Medical University of Graz.

ELIGIBILITY:
Inclusion Criteria:

1. Patient scheduled for treatment with Alirocumab in clinical routine (after approval of cost coverage by insurance company)
2. No previous treatment with PCSK9 antibodies
3. Signed informed consent form

Exclusion Criteria:

1. Age of < 18 years
2. Pregnancy (pregnancy test at screening visit)
3. Breast-feeding
4. Impossibility to perform magnetic resonance imaging of the carotid artery (claustrophobia, carotid stent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Change of mean carotid vessel wall fractional anisotropy (2-Dimensional Cardiovascular Magnet Resonance) by very potent lipid-therapy intensification with Alirocumab | From baseline to 10 weeks of treatment
  Study participants will undergo a cardiovascular magnetic resonance imaging of the carotid vessels. High resolution diffusion tensor imaging (DTI) will be performed on one selected axial slice using read-out segmented EPI (rs-EPI) sequence on a 3T MR scanner.

SECONDARY OUTCOMES:
Change of FDD (flow-dependent dilation) in response to Alirocumab | From baseline to 10 weeks of treatment
  Vasodilation of the brachial artery will be measured with a linear array transducer, 8-13 MHz. Flow mediated dilatation is defined as the change in post-ischemic diameter as a percentage of the baseline diameter. Flow-independent vasodilatation will be evaluated by nitroglycerin-mediated dilatation. At least 15 minutes after the flow mediated procedure the brachial arterial diameter will be measured before and 3 minutes after sublingual administration of nitroglycerin (NTG 0.3 mg spray).
Change of intima media thickness in response to Alirocumab | From baseline to 10 weeks of treatment
  All ultrasound investigations will be performed at the Division of Angiology, Department of Internal Medicine, Medical University of Graz. Carotid intima-media thickness is defined as the mean of at least three different measurements of intima media thickness in a one-centimeter-long segment of the brachial common carotid artery.
Change of post-prandial lipaemia in response to Alirocumab | From baseline to 10 weeks of treatment
  Post-prandial lipaemia will be assessed with a fat-tolerance test (FTT). The participants will receive a standard fat rich meal. The Lipotest® meal is a diagnostic meal with special medical purpose, characterized as "Food for specialized diagnostic determination of postprandial triglycerides" and consists of 832 kCal total energy input (75 g saturated fat, 25 g carbohydrates, 10 g protein, 2,1 g fiber and 0,15 g salt).
Change of the lipoprotein subfractions in response to Alirocumab | From baseline to 10 weeks of treatment
  LDL-Cholesterol will not only be calculated via Friedewald formula, but all plasma lipoprotein particles will be subfractionated by ultracentrifugation / precipitation (Chylomicrons, VLDL, LDL and HDL). Plasma lipid levels will be measured enzymatically using an autoanalyzer. Particle concentrations of lipoprotein subclasses will be measured using nuclear magnetic resonance as previously described (Silbernagel et al 2017). The Apo(lipo)protein levels will be measured using immunoassays.
Changes of inflammatory parameters in response to Alirocumab | From baseline to 10 weeks of treatment
  Enzyme-linked immunosorbent assay kits will be used and C-reactive protein, as well as cytokines and adhesion molecules of special interest.

CONTACTS AND LOCATIONS:
Overall Officials: Günther Silbernagel, MD. Ass.Prof., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No